CLINICAL TRIAL: NCT06874283
Title: Registry and Biobank of Patients With a History of Cancer Therapy
Brief Title: Ocular Complications From Cancer Therapy - Patient Registry and Biobank
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Maryland, Baltimore (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: 24105GCCC
Record Dates: First submitted 2025-02-07; First posted 2025-03-13 (Actual); Last update posted 2025-07-03 (Actual); Status verified 2025-07

CONDITIONS: Graft Versus Host Disease in Eye; Ocular Complications; Inflammatory Dry Eye Disease
Keywords: ocular graft versus host disease; allogenic stem cell transplant; blood cancer; ocular complications; inflammatory dry eye disease; ocular surface disease
MeSH Terms: conditions — Hematologic Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Cancer Therapy (Experimental): The intervention administered will be the eye exam and research protocols (e.g. tear collection, impression cytology, and blood collection)
  Interventions: Procedure: Eye exam
- Control (Active Comparator): The intervention administered will be the standard of care procedures of the eye exam.
  Interventions: Procedure: Eye exam

INTERVENTIONS:
Procedure: Eye exam — Previous medications, ocular history, medical history, clinical evaluations, surgical procedures and outcomes will be gathered on the patients who consent to participate. A standard of care exam will be performed to the reason for the visit. In addition to the standard of care exam, those in the Cancer Therapy arm will have certain biological samples (tear collection, impression cytology, and/or blood) collected, stored, and analyzed so we may obtain immunologic, cellular, or molecular mechanistic insights into disease pathogenesis.

SUMMARY:
The purpose of this study is to collect data on patients seen at University of Maryland after undergoing cancer therapy. Previous medications, ocular history, medical history, clinical evaluations, surgical procedures and outcomes will be gathered on the patients who consent to participate. Potential subjects will be enrolled from the clinical practice of the investigator at the time of their eye examination visit. A standard of care exam will be performed pertinent to the reason for the visit. In addition to the standard of care exam, certain biological specimens (ocular surface wash, mucocellular material, corneal filaments, impression cytology, and/or blood) will be collected, stored, and analyzed to obtain immunologic, cellular, or molecular mechanistic insights into disease pathogenesis.

DETAILED DESCRIPTION:
The objective of this study is to evaluate and study the immunologic changes in patients who undergo cancer therapy, specifically identifying patients who are at risk of developing ocular complications from their cancer therapy such as ocular GVHD and corneal toxicity. By creating a detailed registry and robust biobank of patients' samples, the investigators will have the ability to (1) better define the pathogenesis of the ocular toxicity such as ocular GVHD or corneal keratopathy from cancer immunologics, (2) identify predictive factors for developing ocular complications as a result of cancer therapy. By developing a biobank of patients' samples who have undergone cancer therapy, the investigators will have the ability to evaluate clinical findings and determine factors and markers to better understand the mechanisms corneal disease in these patients. Through this biobank, the investigators would like to gather data on the clinical findings and management of ocular complications in patients who have undergone cancer treatment. Participants will fall into one of two groups: either the the Bone Marrow Transplant/Cancer Therapy group or Control group where they have no previous history of cancer therapy. The intervention in this study will be the eye exam.

ELIGIBILITY:
Inclusion Criteria for the Cancer Therapy Group:

* Adult patients (greater than 18 years of age)
* Deny a history of eye diseases (excluding cataract, glaucoma, mild dry eye disease, or history of cataract or refractive surgery)
* Patients who have a history of allogenic HSCT with all stem cell sources including bone marrow, PBSC, cord AND/OR patients with a history of prior cancer therapy including BMT, chemotherapy, and immunotherapy
* Patients will be recruited after their HSCT or cancer therapy at their ophthalmology appointment
* Patients can be included with a history of prior cancer therapy including chemotherapy, BMT, immunotherapy. Prior cancer therapy must be identified and documented.
* The patient must be able to understand and sign and date the informed consent form approved by the IRB.

Inclusion Criteria for the Control Group:

* No history of cancer or cancer therapy in the past
* Adult patients (greater than 18 years of age)
* Deny a history of eye diseases (excluding cataract, glaucoma, mild dry eye disease, or history of cataract or refractive surgery)
* The patient must be able to understand and sign and date the informed consent form approved by the IRB.

Exclusion Criteria for the Cancer Therapy Group:

* Vulnerable populations: neonates, children, prisoners, institutionalized individuals
* Inability or refusal to provide informed consent.
* History of ocular surgery or ocular disease (except refractive or cataract surgery, mild dry eye disease, or glaucoma).

Exclusion Criteria for the Control Group:

* Vulnerable populations: neonates, children, prisoners, institutionalized individuals
* Inability or refusal to provide informed consent.
* History of ocular surgery or ocular disease (except refractive or cataract surgery, mild dry eye disease, or glaucoma).
* History of cancer or cancer therapy including chemotherapy, immunotherapy, BMT.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 150 (Estimated)
Dates: Start 2025-05-13 (Actual); Primary Completion 2031-04 (Estimated); Study Completion 2031-04 (Estimated)

PRIMARY OUTCOMES:
International Chronic Ocular Graft Versus Host Disease Severity Score | At the time of intervention (eye exam), between on average 3 months to 5 years post-transplant, but this can also extend up to 10 years post-transplant. The expected average will be 3 years post-transplant.
  The International Chronic oGVHD severity score (Ogawa, Y. et al. International Chronic Ocular Graft-vs-Host-Disease (GVHD) Consensus Group: Proposed Diagnostic Criteria for Chronic GVHD (Part I). Sci Rep 3, 3419 (2013). https://doi.org/10.1038/srep03419) is the standard of care for diagnosing and monitoring ocular GvHD. Briefly, this is calculated based on the sum of the patient's Schirmer's severity score (range of 0-3), OSDI severity score (range of 0-3), corneal fluorescein staining severity score (range of 0-3), and conjunctival injection severity score (range of 0-2). This sum ranges from 0 to 11. To diagnose whether a patient has no oGVHD, probable oGVHD, or definite oGVHD, there are two separate scales depending on whether the patient has systemic GVHD or not. Based on the sum of the characteristics, one can diagnose whether or not the patient has oGVHD. Patients are categorized into None, Probable or Definite and the criteria is different based on their systemic GvHD status.

CONTACTS AND LOCATIONS:
Locations (1):
- Stoler Outpatient Cancer Center at the University of Maryland, Baltimore, Maryland, United States

IPD SHARING:
Plan to Share IPD: No